CLINICAL TRIAL: NCT02587481
Title: Pneumological Phenotyping of Acute Coronary Syndrom (ACS) Patients Concerning Concomitant Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Pneumological Acute Coronary Syndrom (ACS) Phenotyping Aachen
Acronym: PAPA
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 15-057
Record Dates: First submitted 2015-10-15; First posted 2015-10-27 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Acute Coronary Syndrom; Chronic Obstructive Pulmonary Syndrom
Keywords: Acute coronary syndrom; Chronic obstructive pulmonary disease; Myocardial infarction; Blood based biomarkers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Blood plasm
Oversight: Data Monitoring Committee: No

SUMMARY:
In this open, monocentric, observational study acute coronary syndrom (ACS) patients will be characterized by pneumological examination concerning a concomitant chronic obstructive pulmonary disease (COPD). Often COPD coexists with ACS; therefore ACS patients benefit either from prevention or potential therapy of chronic hypoxia.

DETAILED DESCRIPTION:
In this study patients with either non ST-segment-elevation myocardial infarction (NSTEMI) or ST-segment-elevation myocardial infarction (STEMI) will be included. After amnesis patients will undergo blood withdrawal, blood-gas analysis and examinations concerning pulmonary function (Bodyplethysmography). In addition to routine blood withdrawal for differential blood count, 9 ml blood sample is takenfor molecular analysis of relevant prognostic chronic obstructive pulmonary disease (COPD)-blood based biomarkers, an for establishing a library of biomaterial in form of a biobank.

ELIGIBILITY:
Inclusion Criteria:

* Written declaration of consent
* Patients with acute myocardial infarct which can be either non ST-segment-elevation myocardial infarct (NSTEMI) or ST-segment-elevation myocardial infarct (STEMI), in both cases exaggeration of cardiac ischaemic markers

Exclusion Criteria:

* Patients not fulfilling the incluson criterias or:
* Pregnant or breastfeeding women
* Participation in other studies
* Persons in depency from the sponsor or working with the sponsor
* Persons without mental ability or capacity to understand and follow the instructions of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with either non ST-segment-elevation myocardial infarction (NSTEMI) or ST-segment-elevation myocardial infarction (STEMI)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with Acute Coronary Syndrom (ACS) and concomitant Chronic Obstructive Pulmonary Disease (COPD) | During 1-2 hours (at time of examination)

SECONDARY OUTCOMES:
Molecular analysis of relevant blood based chronic obstructive pulmonary disease (COPD) biomarkers | An average of 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dreher, Univ.-Prof. Dr. med., Principal Investigator — RWTH Aachen University Hospital MK1; VIncent Brandenburg, apl. Prof. Dr. med, Principal Investigator — RWTH Aachen University Hospital MK1; Christian Cornelissen, Dr. med, Principal Investigator — RWTH Aachen University Hospital MK1
Locations (1):
- Amrei Pelzer, Aachen, North Rhine-Westphalia, Germany